CLINICAL TRIAL: NCT00314990
Title: Homocysteine Lowering by B Vitamins and the Secondary Prevention of Deep-Vein Thrombosis and Pulmonary Embolism. A Randomized, Placebo-Controlled, Double Blind Trial.
Brief Title: VITRO-Trial. B Vitamins and the Secondary Prevention of Venous Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Netherlands Heart Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NHS94.141; NHS99.055
Record Dates: First submitted 2006-04-14; First posted 2006-04-17 (Estimated); Last update posted 2006-04-17 (Estimated); Status verified 2006-04

CONDITIONS: Deep-Vein Thrombosis; Pulmonary Embolism
Keywords: Venous thrombosis; Deep-vein thrombosis; Pulmonary embolism; Homocysteine; B-vitamins; Folate; Vitamin B12; Vitamin B6
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Folic Acid; Pyridoxine; Vitamin B 12

INTERVENTIONS:
Drug: 5 mg folic acid, 50 mg pyridoxine and 0.4 mg cyanocobalamin

SUMMARY:
The VITRO (Vitamins and Thrombosis) study investigated the effect of homocysteine lowering by daily supplementation of B-vitamins on the risk reduction of deep-vein thrombosis and pulmonary embolism. Patients between 20 to 80 years old with a first objectively confirmed proximal deep-vein thrombosis or pulmonary embolism in the absence of major risk factors and a homocysteine concentration above the 75th percentile of a reference group were asked to participate (hyperhomocysteinemic group). A similar study was conducted in a random sample of patients with a homocysteine below the 75th percentile of the reference group (normohomocysteinemic group). After informed consent patients were randomized to daily multivitamin supplementation (5 mg folic acid, 50 mg pyridoxine and 0.4 mg cyanocobalamin) or placebo and were followed for 2.5 years. End-points were objectively diagnosed recurrent deep-vein thrombosis or pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* objectively confirmed proximal deep-vein thrombosis or pulmonary embolism
* idiopathic thrombosis (i.e. absence of major risk factors (major surgery, known malignant disease, pregnancy and puerperium or immobility for more than three weeks)
* age between 20 to 80 years

Exclusion Criteria:

* obligatory use of vitamin B

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620
Dates: Start 1996-01; Study Completion 2003-01

PRIMARY OUTCOMES:
Recurrent symptomatic DVT or recurrent PE.

CONTACTS AND LOCATIONS:
Overall Officials: Martin den Heijer, MD PhD, Principal Investigator — Radboud University Medical Center; Gerard MJ Bos, MD PhD, Study Director — Maastricht University Medical Center
Locations (1):
- Leyenburg Hospital (currently HAGA-hospital), The Hague, Netherlands

REFERENCES:
- [Derived] den Heijer M, Willems HP, Blom HJ, Gerrits WB, Cattaneo M, Eichinger S, Rosendaal FR, Bos GM. Homocysteine lowering by B vitamins and the secondary prevention of deep vein thrombosis and pulmonary embolism: A randomized, placebo-controlled, double-blind trial. Blood. 2007 Jan 1;109(1):139-44. doi: 10.1182/blood-2006-04-014654. Epub 2006 Sep 7. PMID 16960155